CLINICAL TRIAL: NCT05471219
Title: THE EFFECT OF FOCUS APPLICATION DURING THE FIRST VAGINAL EXAMINATION IN TRAVEL ON THE VAGINAL EXAMINATION EXPERIENCE AND PAIN LEVEL OF PREGNANT PREGNANCY: A RANDOMIZED CONTROLLED STUDY
Brief Title: The Effect of Focus on Vaginal Examination Experience and Pain Level: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek Yigit Vural (Other)
Responsible Party: Sponsor-Investigator, Dilek Yigit Vural, Midwife, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D.2021-2022
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Birth, First; Experience, Life; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Çalışma grubu (Experimental): Primiparous pregnant women who will undergo vaginal examination by focusing on visual traces
  Interventions: Other: Primiparous pregnant women who will undergo vaginal examination by focusing on visual traces
- Kontrol grubu (No Intervention): Primiparous pregnant women who will undergo vaginal examination with standard care

INTERVENTIONS:
Other: Primiparous pregnant women who will undergo vaginal examination by focusing on visual traces — Informed consent was obtained from the mothers to take pictures of newborns who were delivered in the delivery room, routinely cared for, dressed and breastfed by the researcher. A 10-minute visual track was created to be turned into a slide from approximately 70 photos. Vaginal examination was performed between the 4th and 6th minutes while focusing on this visual trace.
  Arms: Çalışma grubu

SUMMARY:
Vaginal examination contains many negative emotions such as pain, fear, stress, and discomfort for women. When the literature was examined, no study was found in which the focus method was used to reduce or eliminate the feelings that cause negative emotions in women in the vaginal examination experience. For this reason, our research will be a first in the literature and it is thought that it will contribute to the field. In this context, it is assumed that the focusing behavior based on the door control theory will reduce the pain level of primiparous women who will have a vaginal examination for the first time in labor, positively affect the vaginal examination experience and experience a positive birth. In the research; Ho hypothesis: Focus has no effect on the vaginal examination experience of pregnant women.

Hypothesis H1: Focus has an impact on the vaginal examination experience of pregnant women.

Ho hypothesis: Focus has no effect on vaginal examination pain level of pregnant women.

Hypothesis H1: Focus has an effect on the vaginal examination pain level of pregnant women.

It was aimed to examine the effect of focusing on the first vaginal examination experience and pain level of primiparous women in labor by establishing hypotheses.

DETAILED DESCRIPTION:
Vaginal examination before and during labor may cause negative feelings in women and adversely affect the birth. Distraction attempts to be made during the examination process can help the pregnant woman both self-confidence and take the first step towards a positive birth. This study was conducted to examine the effect of the focus applied during the first vaginal examination in labor on the vaginal examination experience and pain level of primiparous pregnant women. The study was conducted in a randomized controlled clinical trial design with primiparous women who applied to give birth in Ankara City Hospital Gynecology clinic between June and November 2021. 102 (study: 51, control: 51) women determined by the G*Power 3.1 program were included in the research sample. Research data were collected through an introductory information form, a visual comparison scale, and a scale of women's expressions of vaginal examination in labor. Data were analyzed with IBM SPSS V23. Compliance with normal distribution was examined by Shapiro-Wilk and Kolmogorov-Smirnov tests, and when comparing normally distributed data in paired groups, independent two-sample t-test was used, and when comparing non-normally distributed data, Mann Whitney U Test was used. One-Way Analysis of Variance was used to compare the normally distributed data in the three groups, the Kruskal Wallis Test was used to compare the non-normally distributed data, and the Chi-Square Test was used to compare the categorical data. Spearman's rho correlation coefficient was used to examine the relationship between non-normally distributed variables and scale scores. Linear Regression Analysis was used to determine the independent variables affecting the scale score and VAS score. The results are presented as frequency (percentage) for categorical variables, mean ± standard deviation and median (minimum - maximum) for quantitative variables.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* The gestational week is due,
* Able to speak and understand Turkish,
* Single and healthy fetus pregnancy,
* Primiparous,
* Head presentation,
* No diagnosis of risky pregnancy,
* Not allergic to latex,
* Having a vaginal examination for the first time after being admitted to the TDL service,
* In the latent phase (examination between 0-5 cm when applying to the emergency department (WHO, 2018))
* No communication problem,
* Does not have a mental illness,
* No premature rupture of membranes,
* Pregnant women who agreed to participate in the study.

Exclusion Criteria:

* Genito-urinary system infection,
* Having vaginismus,
* Pregnant women whose first vaginal examination was not performed by the researcher during labor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 15-minute time frame immediately after the vaginal exam
  It is a scale used to measure perceived pain. In the form of a 0-10 cm ruler, one end of the scale indicates 0 painlessness and the other end 10 indicates the most severe pain intensity degree. The degree of pain intensity was evaluated by marking the perceived pain of the pregnant woman on the ruler.
The Women's Experiences of Vaginal Examinations in Labour Scale | 15-minute time frame immediately after the vaginal exam
  The Vaginal Examination Experiences of Women in Labor Scale is a 5-point Likert-type scale consisting of 20 items. In the scale, 9 items (5, 10, 13, 14, 15, 16, 17, 19 and 20) are reverse scored. The scale consists of five sub-dimensions. For the sub-dimensions of the scale, the scores of the items in each sub-dimension were summed and the raw scores were divided by the number of items, and sub-dimension scores between 1-5 were obtained. These scores are multiplied by 20 to obtain a sub-dimension score between 20-100. A minimum of 20 points and a maximum of 100 points can be obtained from the scale. Accordingly, the higher the score of an item, the more satisfied the participant will be with the vaginal examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital/Gynecology and Obstetrics Hospital, Ankara, Turkey (Türkiye)